CLINICAL TRIAL: NCT00916279
Title: A Prospective, Multicenter, European Registry Investigating the Lutonix Paclitaxel-Coated Balloon for the Treatment of In-Stent Restenosis Within Bare-Metal Stents
Brief Title: PERVIDEO I Registry, The Lutonix Paclitaxel-Coated Balloon Catheter for the Treatment of Coronary In-Stent Restenosis
Acronym: PERVIDEO I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0010-01
Record Dates: First submitted 2009-06-04; First posted 2009-06-09 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: In-Stent Restenosis
Keywords: Bare Metal In-Stent Restenosis; Paclitaxel Coated Balloon Catheter; Drug Coated Balloon; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lutonix Catheter (Experimental)
  Interventions: Device: Lutonix Paclitaxel-Coated Balloon

INTERVENTIONS:
Device: Lutonix Paclitaxel-Coated Balloon — PTCA
  Other Names: Drug Coated Balloon

SUMMARY:
The study will enroll patients with angiographic evidence of in-stent restenosis of a previously placed bare-metal stent. Subjects will be treated with a Lutonix Catheter. The purpose is to investigate the feasibility, safety, and efficacy of the Lutonix Catheter in the native coronary system. Angiographic and clinical outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant/non-breast feeding Female ≥18 Years of age. Women of childbearing potential must have a negative pregnancy test within 7 days of the procedure;
* Documented stable angina pectoris Canadian Cardiovascular Society Classification (CCSC) 1-4, unstable angina pectoris with documented ischemia (Braunwald I-II) or documented silent ischemia;
* Previous history of native coronary bare metal stenting ≥60 days;
* LVEF ≥25%;
* Patient is an acceptable candidate for PTCA, stenting, and emergent CABG;
* Patient is willing to provide informed consent and comply with follow-up visits and testing schedule;
* Target lesion is in a native coronary with previous single bare metal stent; Stenosis is ≥50% and <100% by visual estimate or QCA prior to defined pre-dilatation;
* Reference Vessel Diameter (RVD) is ≥2.5 and ≤3.25;
* Target lesion is ≤40 mm in length and can be treated in its entirety by no more than 2 contiguous Lutonix Catheters;
* Guidewire is able to cross lesion(s) and be placed in distal vessel prior to enrollment;
* Enrollment permitted after successful treatment of 1 to 2 non-study lesions in a single other non-study vessel. Successful treatment is defined as ≤30% residual stenosis with TIMI III flow and no evidence of dissection.

Exclusion Criteria:

* History of Stroke within past 6 months;
* History of MI or thrombolysis within 72 hours of randomization;
* History of previous target vessel perforation;
* Prior vascular brachytherapy;
* Angiographic evidence of thrombus or dissection within the target vessel;
* Intervention of another coronary lesion <60 days before index procedure day or planned following index procedure;
* Target lesion is in the Left Main or vessel ostium and has excessive calcification or tortuosity or involves bifurcation disease of vessel ≥2.5 mm;
* Target lesion is planned to be treated with something other than PTCA (i.e. stent, cutting balloon, atherectomy, VBT, etc.);
* Uncontrollable allergies to procedure medications, materials, or contrast;
* Patient has previous stent procedure with any drug-coated or drug eluting stent device in the target coronary vessel;
* Known sensitivity to paclitaxel or other antimitogenic agent;
* Patient has a stent sandwich (a stench previously deployed within another stent;
* Pre-procedure CKMB >2x ULN or positive Troponin;
* Creatinine >2.0 mg/dl;
* Leukocyte <3500/mL;
* Platelet <100,000 mL or >750,000 mL;
* Currently taking or must resume warfarin;
* Patient is contraindicated for anti-platelet therapy or it will need to be withdrawn for a planned procedure;
* The patient is currently participating in another investigational drug or device study that has not completed its primary endpoint or that clinically interferes with the endpoints of this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mauri, MD, Principal Investigator — Brigham & Women's Hospital, Boston, MA
Locations (8):
- Onze Lieve Vrouw Ziekenhuis, Aalst, Belgium
- Germany (4):
  - Kerckhoff Klinik, Bad Nauheim
  - Westdeutsches Herzzentrum Essen, Essen
  - Alte Clinic Center for Cardiology, Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Catherina Ziekenhuis, Eindhoven
  - Sint Antonius Ziehenhuis, Nieuwegein

REFERENCES:
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Speck U, Scheller B, Abramjuk C, Breitwieser C, Dobberstein J, Boehm M, Hamm B. Neointima inhibition: comparison of effectiveness of non-stent-based local drug delivery and a drug-eluting stent in porcine coronary arteries. Radiology. 2006 Aug;240(2):411-8. doi: 10.1148/radiol.2402051248. PMID 16864669
- [Background] Stone GW, Ellis SG, O'Shaughnessy CD, Martin SL, Satler L, McGarry T, Turco MA, Kereiakes DJ, Kelley L, Popma JJ, Russell ME; TAXUS V ISR Investigators. Paclitaxel-eluting stents vs vascular brachytherapy for in-stent restenosis within bare-metal stents: the TAXUS V ISR randomized trial. JAMA. 2006 Mar 15;295(11):1253-63. doi: 10.1001/jama.295.11.1253. Epub 2006 Mar 12. PMID 16531618
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Holmes DR Jr, Teirstein P, Satler L, Sketch M, O'Malley J, Popma JJ, Kuntz RE, Fitzgerald PJ, Wang H, Caramanica E, Cohen SA; SISR Investigators. Sirolimus-eluting stents vs vascular brachytherapy for in-stent restenosis within bare-metal stents: the SISR randomized trial. JAMA. 2006 Mar 15;295(11):1264-73. doi: 10.1001/jama.295.11.1264. Epub 2006 Mar 12. PMID 16531619
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Kastrati A, Mehilli J, von Beckerath N, Dibra A, Hausleiter J, Pache J, Schuhlen H, Schmitt C, Dirschinger J, Schomig A; ISAR-DESIRE Study Investigators. Sirolimus-eluting stent or paclitaxel-eluting stent vs balloon angioplasty for prevention of recurrences in patients with coronary in-stent restenosis: a randomized controlled trial. JAMA. 2005 Jan 12;293(2):165-71. doi: 10.1001/jama.293.2.165. PMID 15644543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from June 3, 2009 through December 8, 2009 at 7 centers in Germany, Netherlands, and Belgium.
Groups:
- Lutonix DCB Catheter: Lutonix Paclitaxel-Coated Balloon: PTCA
Period: Overall Study
Arm/Group | Lutonix DCB Catheter
Started | 41
30 Days | 41
6 Months | 41
24 Months | 37
Completed | 37
Not Completed | 4
Not completed — Death | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lutonix Catheter
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (11.0)
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 31
Region of Enrollment [Number; unit: participants]
  Belgium | 1
  Netherlands | 4
  Germany | 36
Target Lesion Location [Number; unit: participants] — Target coronary vessel(s) treated: circumflex (CFX), left anterior descending (LAD), right coronary artery (RCA).
  participants
    CFX | 17
    LAD | 13
    RCA | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Diameter Stenosis (%DS) in the Analysis Segment
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: Percentage stenosis of vessel diameter
Groups:
- Lutonix DCB Catheter: Lutonix paclitaxel-coated PTCA balloon catheter
Arm/Group | Lutonix DCB Catheter
Number analyzed (Participants) | 41
Percentage stenosis of vessel diameter | 36.0 (17.6)

2. Secondary Outcome: Late Lumen Loss
Description: Change in (loss of) lumen diameter from baseline through 6 months in the analysis segment (including the treated segment and 5mm proximal and distal).
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: (mm)
Arm/Group | Lutonix Catheter
Number analyzed (Participants) | 41
(mm) | 0.17 (0.39)

3. Secondary Outcome: MACE Rate
Description: Major adverse coronary events (MACE), including the composite of cardiac death, myocardial infarction (MI), and target vessel revascularization (TVR).
Time Frame: 30 Days
Population: ITT
Measure: Number; unit: Percentage of patients
Groups:
- Lutonix PTCA Catheter: Lutonix Paclitaxel-Coated Balloon: PTCA
Arm/Group | Lutonix PTCA Catheter
Number analyzed (Participants) | 41
Percentage of patients | 0

4. Primary Outcome: Change in Diameter Stenosis (%DS) From Post-procedure Through 6 Months
Description: Paired change in percent diameter stenosis (%DS) in the analysis segment from post-procedure through 6 months. I.e., %DS at follow-up less %DS post procedure per patient.
Time Frame: 6 Months
Population: ITT
Measure: Mean (Standard Deviation); unit: percent diameter stenosis
Arm/Group | Lutonix DCB Catheter
Number analyzed (Participants) | 41
percent diameter stenosis | 8.5 (16.9)

5. Secondary Outcome: Binary Restenosis
Description: Subjects with percent diameter stenosis >50% in the analysis segment.
Time Frame: 6 Months
Population: ITT
Measure: Number; unit: participants
Arm/Group | Lutonix DCB Catheter
Number analyzed (Participants) | 41
participants | 5

ADVERSE EVENTS:
Arm/Group | Lutonix Catheter
Serious Adverse Events (participants affected / at risk) | 22/41
Other Adverse Events (participants affected / at risk) | 15/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix Catheter (N=41)
Death of unknown cause (Injury, poisoning and procedural complications) | 1 (1)
Abdominal aortic aneurysm (Injury, poisoning and procedural complications) | 1 (1)
Acute renal failure post-interventional (Renal and urinary disorders) | 1 (1)
Rotoblation of non-target vessel/fell into lung edema & ventricular fibrillation. Resulted in death (Injury, poisoning and procedural complications) | 1 (1)
Aneurysm spurium of RCA (Injury, poisoning and procedural complications) | 1 (1)
Aneurysma rupture by distal endoleak right iliacal (Injury, poisoning and procedural complications) | 1 (1)
Angina (Cardiac disorders) | 6 (8)
Bacteria MIC = staphylococcus auras (Infections and infestations) | 1 (1)
Cardiac decomposition with pneumonia and sepsis and respiratory insufficiency due to pulmonary edema (Cardiac disorders) | 1 (1)
CCSIII caused angio. Occlusion of prox. RCA NTVR done (Cardiac disorders) | 1 (1)
Effective reconstruction: RCA - 3 DES stents (atypical chest pain / discomfort, angiographic stenosi (Cardiac disorders) | 1 (1)
Hospitalization (General disorders) | 2 (2)
Hypertensive Crisis (Renal and urinary disorders) | 1 (1)
Instent Restenosis (Vascular disorders) | 2 (2)
Kidney Stones (Renal and urinary disorders) | 1 (1)
Nasal bleeding / epistaxis (General disorders) | 1 (1)
Dyspnea and Thorax Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial abscess (Cardiac disorders) | 1 (1)
Perimyocarditis with pericardial effusion (Cardiac disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Progression of coronary artery disease proximal to treated lesion (non-TLR-PCI) (Cardiac disorders) | 1 (1)
Recurrent Depressive disorder, pre-existing condition (Psychiatric disorders) | 1 (1)
Reintervention (Injury, poisoning and procedural complications) | 1 (1)
Re-PCI (Cardiac disorders) | 2 (2)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Stenosis (Vascular disorders) | 4 (5)
Thoracic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix Catheter (N=41)
Angina (Cardiac disorders) | 6 (6)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypertension (Renal and urinary disorders) | 7 (7)
Palpitations (Cardiac disorders) | 2 (3)
Thoracic Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other